CLINICAL TRIAL: NCT05158712
Title: Genetic Modifying Factors and Pheochromocytomas in Multiple Endocrine Neoplasia Type 2
Brief Title: Genetic Factors and Pheochromocytomas in Neoplasia Type 2
Acronym: NEM2A-Pheo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-65
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Neoplasia; Pheochromocytoma
Keywords: neoplasia; pheochromocytoma
MeSH Terms: conditions — Neoplasms; Pheochromocytoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple endocrine neoplasia type 2A (MEN2A) is a rare syndrome associated with activating mutations in the RET proto-oncogene, combining medullary thyroid cancer in approximately 100% of cases and pheochromocytoma in 10-80% of cases. While it is accepted that the RET mutation causes variable penetrance of pheochromocytoma in the MEN2A patient population, there is no pathophysiological explanation for the phenotypic variability among patients with the same mutation, including within the same family. The aim of this study is to better characterise the genetic factors that may explain the variable penetrance of pheochromocytoma in MEN2. To this end, the investigatoes plan to perform a whole exome analysis in 2 families carrying the p. Cys634Arg mutation causing NEM2A, followed in Marseille by the principal investigator: the 1st family has 11 members all aged over 35 years, for which 8 are carriers of pheochromocytoma while 3 have not developed it (while their age is higher than the latest age of diagnosis of pheochromocytoma in this family); the 2nd family has 3 members (father and daughter with pheochromocytoma developed before 25 years; son without pheochromocytoma at an age of 42 years). The investigators believe that the analysis of these patients should allow the isolation of variants on genes potentially involved in the genesis of a pheochromocytoma in MEN2.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Male or female patient
* Patient followed in the investigating department for familial NEM2A C634R (multiple endocrine neoplasia type 2) with or without pheochromocytoma
* Patient affiliated to or benefiting from a social security scheme
* Patient having given his non-opposition to participate in this study
* Patient who has given his consent for the genetic analysis carried out in the framework of the study
* Patient able to understand the purpose of the study

Exclusion Criteria:

* Protected persons (articles L1121-5, L1121-6 and L121-8 of the Public Health Code): pregnant or breastfeeding women, persons deprived of their liberty, under guardianship or curator
* Patients unable to understand the purpose of the study and the information note

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient followed for familial neoplasia type 2 with or without pheochromocytoma
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Genetic profile | Month 0
  whole-exome analysis between patients with and without pheochromocytoma

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — APHM
Locations (1):
- APHM - Hôpital de la Conception, Marseille, France

IPD SHARING:
Plan to Share IPD: No